CLINICAL TRIAL: NCT06496464
Title: Professor Dr Jin Yan (PhD in Education)
Brief Title: We Designed and Implemented the 'MASTER Framework' as a Theoretical Framework to Guide the Design and Delivery of PE and Sports.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Soochow University (Other)
Responsible Party: Principal Investigator, Jin Yan, Pro Dr, Soochow University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SUDA20240626H06
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Help PE Teachers Learn and Develop the Critical Skills Needed to Create a Positive Teaching Environment
Keywords: Teaching; sport; Education; motivation; well-being; game-based approach
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: The MASTER teacher education program is developed and designed based on the findings of a pilot study by the research team at the University of Newcastle. The basis of MASTER is the so-called "positive teaching", and the concept is fostered and promoted through the teaching practices based on the games; its targets include six critical sports teaching elements, which are proven to promote well-being, health, and physical outcomes in children. Eather, Jones, et al. (2020) have demonstrated that PE teachers try to make use of the MASTER framework, which is not only user-friendly but also evidence-based, as a practical instrument when planning and delivering sessions of soccer training with high quality, which meets the interests of children such as exercise, teamwork, skill development, and success, and helps the children to improve learning and give full play to the potential.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): Teachers randomized to the control group will participate in the following:
  Basketball training as usual, which involves one 2-3 hour session delivered per week based on local school protocol
  Teachers in the control group will only receive the MASTER Teaching Program after completing the study period and assessing outcome measures.
  Interventions: Behavioral: Intervention
- Intervention condition (MASTER teacher education program) (Experimental): Jin Yan will train the PE teachers to complete video assessments and questionnaires. Five teachers from the intervention group will be educated in the MASTER coach education program and trained to deliver a basketball program that aligns with the MASTER framework.
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Phase 1 MASTER Coach Development Workshop (weeks 1) PE teachers participated in a 6-hour theory and practical teacher education workshop to a research team (JY) member, including 4h of reading relevant papers and books regarding the game-based approach (GBA) .
  Phase 2 Eight weeks of teaching mentoring (weeks 2-7) This 8-week phase involved coaches implementing MASTER elements (e.g. 10-minute stretching before a sports game, teachers will give 1-2 sentences of praise during the game for individual students who make a reasonable effort) in their regular training sessions.
  Phase 3 3 weeks peer assessed teaching/discussions (weeks 8-10) The mentor prepared and implement a 2-h training session designed to highlight important aspects of the MASTER framework and games-based coaching practices.

SUMMARY:
Our research team is committed to improving the quality of physical education in China. Based on the needs of teachers and sports coaches in China, we designed and implemented the 'MASTER Framework' as a theoretical framework to guide the design and delivery of PE and sports. This framework aims to help PE teachers learn about and develop the critical skills needed to create a positive teaching environment and facilitate effective PE class delivery using a games-based approach (GBA).

DETAILED DESCRIPTION:
Phase 1 MASTER Coach Development Workshop (weeks 1) PE teachers participated in a 6-hour theory and practical teacher education workshop via Zoom to a member of the research team (JY), including four hours of reading relevant papers and books regarding the game-based approach (GBA) (Game-sense, Invasion Games, Small-sided games and tactical approach). The latest evidence regarding sport, coaching and youth was presented, and the MASTER framework was explained. A combination of lectures, discussions and group work activities provided coaches with the theoretical underpinnings and practical applications of the MASTER elements. It allowed coaches to plan and assess sessions based on the MASTER framework and evaluation tool. A key target for the workshop was to empower coaches with the necessary skills and understanding to use the MASTER framework when designing new training activities or adapting existing activities. Coaches were provided with a PowerPoint presentation, printed course booklet, MASTER checklist, and printed (and explained) examples of basketball training activities and planning tasks. The workshop components (e.g., PowerPoint presentations, workshop materials, practical sessions) were designed and developed to minimise the impact of the presenters' biographies on knowledge uptake and ensure suitability for future scale-up (whereby external presenters would deliver the MASTER program).

Phase 2 Eight weeks of teaching mentoring (weeks 2-7) This 8-week phase involved coaches implementing MASTER elements (e.g. 10-minute stretching before a sports game, teachers will give 1-2 sentences of praise during the game for individual students who make a reasonable effort) in their regular training sessions (2 x 1 ½ hour sessions per week) under the guidance of the coach mentor (2-3 experienced coaches who from the member of the research team will evaluate the mentor). The mentor spent one session per week (1 ½ hour) for eight weeks, rotating between coaches to assist in applying the MASTER framework and providing ongoing support. This included access to a discussion platform on Facebook messenger, providing example session activities and MASTER learning activities via the purpose-designed MASTER website, and feedback on draft session plans. During and after the training sessions, the mentor also stimulated dialogue and provided input to coaches regarding potential ways to increase the engagement of players (e.g., adaption of the session activities), questioning techniques to facilitate player reflection and learning, session evaluation and coach reflection; identification of the elements of MASTER in action; and identification of the potential missed opportunity to include an element of MASTER.

Phase 3 3 weeks peer peer-assessed teaching/discussions (weeks 8-10) The mentor prepared and implemented a 2-hour training session highlighting important aspects of the MASTER framework and games-based coaching practices. Coaches were involved in evaluating the mentor using the MASTER observation checklist, and a group discussion based on the checklist and coach observations facilitated the learning episode. This collaborative practise incorporates what is known about professional learning communities and instructional "rounds", and is now common in higher educational settings. The literature supports that learning and understanding are optimised when learners are involved in the feedback process, explicitly learn to become assessors, have a clear framework to evaluate performance, and provide feedback through a discussion or dialogue. Following the coach assessment and reflection session, coaches continued implementing MASTER strategies in their regular training sessions. They were required to undertake a peer observation of a colleague alongside the coach mentor (using the MASTER observation checklist). Feedback and professional dialogue followed the peer observation sessions. Peer dialogue has shown to be an effective and well-received method for improving coaching practices.

Frequency: Participated teachers will be asked to participate in Weekly 2-3 hour game sessions in school, which is an additional component of the intervention (with the teacher's regular class). The sessions will be facilitated by the teacher and supervised by a study team member (weekly 30-40-minute telephone calls with members of the research team discussing strategies for improving game sessions).

ELIGIBILITY:
Inclusion Criteria:

* Only participants providing signed consent were eligible to participate in the study and complete the teacher, student or parent questionnaire.

Exclusion Criteria:

* without an illness or injury that would preclude them from participating in physical activity.

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
PE teacher Confidence and Competence | 2 weeks
  PE Teacher questionnaire: PE teachers will be also asked to complete a purpose-designed questionnaire collecting 1) Confidence to teach basketball; 2) Competence to teach basketball. The teachers' Confidence to teach basketball and Competence to teach basketball will be analysed together as a composite outcome.
Student assessments | 2 weeks
  Students' game skills (assessed at Basketball lesson): Video analysis of decision-making, and attacking and defensive play will be conducted using a previously validated game performance assessment instrument (Miller et al., 2015). These skills are deemed essential for success in invasion games (including basketball) and are skills utilised by all players on the court (irrespective of position played).

SECONDARY OUTCOMES:
Student perceptions | 2 weeks
  Student assessments: Enjoyment of Sport (Basketball Lesson). It will be using an adapted version of the Physical Activity Children's Enjoyment.